CLINICAL TRIAL: NCT05795088
Title: Role of Continuous Theta Burst Stimulation as Potential Biomarker of Levodopa-induced Dyskinesias in Patients With Parkinson's Disease.
Brief Title: Continuous Theta Burst Stimulation as Potential Biomarker of Levodopa-induced Dyskinesias in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 3884
Record Dates: First submitted 2023-02-21; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with parkinson's disease (Experimental)
  Interventions: Device: Continuous theta burst stimulation

INTERVENTIONS:
Device: Continuous theta burst stimulation — Two sessions of continuous theta burst stimulation over primary motor cortex to explore synaptic plasticity in Patients with Parkinson's disease

SUMMARY:
The primary endpoint of the study is to identify a neurophysiological biomarker (absence of synaptic depotentiation at primary motor cortex , measured as change in the amplitude of motor evoked potentials recorded at the dorsal first interosseus muscle after administration of neurophysiological cTBS depotentiation protocol) as predictor of the development of Levodopa-induced dyskinesia in patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* patients with diagnosis of idiopathic Parkinson's disease according to Movement Disorder Society (MDS) criteria;
* age between 30 and 80 years;
* ongoing therapy with levodopa;
* fulfillment of requirements for the application of transcranial magnetic stimulation (TMS), assessed by completion of the TMS screening questionnaire.

Exclusion Criteria:

* patients unable to give informed consent;
* cognitive impairment (MMSE ≤ 24);
* history of epilepsy;
* pregnant women.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-16 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Alterations of synaptic depotentiation in primary motor cortex | 3 years
  Alterations of synaptic depotentiation in primary motor cortex will be measured as change in the amplitude of motor evoked potentials recorded at the dorsal first interosseus muscle after administration of depotentiation protocol of continuous theta burst stimulation. Alterations of synaptic depotentiation at the baseline evaluation will be compared between patients who will develop and patients who will not develop dyskinesias (assessed by Unified Dyskinesia Rating Scale part III, range 0-112) during the follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Calabresi, MD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Flavia Torlizzi, Rome, Italy